CLINICAL TRIAL: NCT03092505
Title: Herpesviruses Reactivation In Hiv-Infected Women Initiating ART (HERA)
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 170072; 17-I-0072
Record Dates: First submitted 2017-03-22; First posted 2017-03-28 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-08-12

CONDITIONS: Herpes Virus-Related Illnesses
Keywords: HSV; Uganda; Sample; Natural History

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Females: Females participants who are about to start first line antiretroviral therapy.

SUMMARY:
Background:

Herpes virus can cause sores on the body. It can cause flu-like symptoms like fever and muscle aches, and even a type of cancer. Many people with HIV also have infections with herpes virus. When these people start taking HIV medicines, their herpes virus symptoms can suddenly start or become worse. Researchers want to find out more about how often this happens and why.

Objective:

To study the effects of HIV treatment in women who may have herpes virus infections.

Eligibility:

Women age 18 years and older who have been diagnosed with HIV infection.

Design:

Participants will be screened with a physical exam, medical history, and blood and urine tests.

Participants will have about 8 study visits. Each will take about 1-2 hours.

Participants will return to the clinic 1-2 weeks after the screening visit to receive their antiretroviral (ART) medicine. They will get instructions for taking it.

Participants will have 6 more study visits over 1 year.

During study visits, participants will have blood and urine tests, vaginal fluid collected, and an oral swab. They may have an external genital exam. They will get their next supply of ART medicine.

Some participants may have a chest x-ray.

Participants may have leukapheresis. Blood will be removed through a needle in an arm. It will be run through a machine that separates out the white blood cells. The rest of the blood will be returned through a needle in the other arm.

The total time participants will be in the study is about 1 year.

DETAILED DESCRIPTION:
Initiation of antiretroviral therapy (ART) can lead to a short-term increase of herpes virus-related illnesses including genital herpes flares, higher likelihood of varicella zoster virus (VZV), cytomegalovirus (CMV) uveitis or other end-organ disease, and herpes simplex virus (HSV) associated encephalitis. Herpesvirus reactivation upon ART initiation may be related to immune restoration disease of immune reconstitution inflammatory syndrome (IRIS), but the etiology is unclear. We hypothesize that ART initiation can induce herpesvirus reactivation causing increased cellular, systemic, and localized immune activation and that alterations of interferon (IFN) pathways during initial HIV viral suppression are involved in this reactivation.

To investigate these mechanisms, we propose to document the incidence of clinical herpetic disease and viral shedding in vaginal and oral secretions from HIV-positive women initiating ART and to assess the associations between viral shedding or clinical disease and cellular, mucosal, and systemic immune activation. We will determine the role of IFN pathway in herpesvirus reactivation following initiation of ART. We will also evaluate the potential impact of herpesvirus reactivation on HIV cellular reservoirs by comparing residual HIV plasma viral replication and cell-associated virus prior to and 52 weeks after ART initiation.

We propose to enroll up to 200 HIV-infected women initiating ART at the NIH Clinical Center (n=30 to 40) and between the Villa Maria Hospital, Rakai Health Sciences Program (RHSP) site in Kalisizo, Uganda and Kalisizo Hospital ARV clinic (n=160 to 170). Women will be recruited regardless of CD4+ T-cell count, presence of opportunistic infections and co-infection status. Pregnant women will be excluded. During 8 study visits to occur over a 12-month period, participants will receive standard-of-care treatment for HIV and opportunistic infections. Blood, vaginal fluid and oral swabs collected at study visits will be tested for viral levels of HIV and various herpesviruses. Vaginal samples will also be used to study differences in vaginal microbiota between women with and without herpetic disease prior and after ART. Plasma samples will be tested for antibody levels (IgG) specific for different herpesviruses to examine changes in anti-herpetic humoral responses. ART adherence will be monitored in plasma using high-resolution mass spectrometry.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. At least 18 years of age
  2. Female
  3. Weight >40 kilograms
  4. A diagnosis of HIV infection as documented by any positive serological test (ELISA, HIV rapid test, or Western Blot)
  5. Participants in Uganda must be eligible for ART by current clinical guidelines in Uganda
  6. Willingness to begin ART
  7. Will allow storage of biological sample

EXCLUSION CRITERIA:

1. Previous exposure to ART (participants with a brief exposure (<3 months) that occurred greater thatn or equal to 6 months prior to screening will be eligible to enroll if, the opinion of the investigator, the ART usage will not impact the scientific validity of the protocol)
2. On acyclovir, valacyclovir, valganciclovir, or ganciclovir treatment
3. Pregnancy or intent to become pregnant during the study period
4. Intrauterine device (IUD) use
5. Inability to follow study instructions, according to the investigator's judgment
6. Active, serious infections other than HIV infection that may interfere with study participation (eg, severe cerebral toxoplasmosis or cryptococcal meningitis) during the 2 weeks prior to enrollment
7. Malignancies requiring chemotherapy
8. Therapy with systemic corticosteroids, immunosuppressants or immunomodulating agents
9. Any condition that, in the investigator s opinion, may put the participant at undue risk or compromise the study's scientific objectives

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 200 women initiating ART as part of standard HIV care will be recruited at four sites, the NIH Clinical Center (approximately 30-40), the RHSP/ICER , the Villa Maria Hospital and the Kalisizo sites in Uganda (approximately 160-170). Women will be recruited regardless of CD4+ T-cell count, presence of opportunistic infections and co-infection status. Participants taking antibiotics for co-infections and prophylaxis will be able to participate in the study and antibiotic use will be captured in study data. Participants may co-enroll in other non-interventional studies. Pregnant women will be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 190 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-04 (Actual)

PRIMARY OUTCOMES:
Compare the prevalence of herpetic disease, demonstrated by viral shedding of HSV-1 and 2 in the vaginal secretions of HIV-positive women prior to and 4 and 8 weeks after ART initiation. | prior to and at 4 and 8 weeks after inititian of antiretroviral treatment
  viral shedding of HSV-1 and 2

SECONDARY OUTCOMES:
1. To estimate the associations of viral shedding or clinical herpetic disease post-ART at weeks 4 or 8 with concurrent and baseline measurement of systemic inflammation (IL-6, CRP, TNF or sCD14). [ Time Frame: 8 weeks post enrollment ] | at week 4 and at week 8

CONTACTS AND LOCATIONS:
Overall Officials: Steven J Reynolds, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (2):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States
- Rakai, Kalisizo, and Villa Maria Hospital, Kalisizo, Uganda

REFERENCES:
- [Background] Schaftenaar E, Verjans GM, Getu S, McIntyre JA, Struthers HE, Osterhaus AD, Peters RP. High seroprevalence of human herpesviruses in HIV-infected individuals attending primary healthcare facilities in rural South Africa. PLoS One. 2014 Jun 10;9(6):e99243. doi: 10.1371/journal.pone.0099243. eCollection 2014. PMID 24914671
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2017-I-0072.html